CLINICAL TRIAL: NCT03561441
Title: Tailored Hydration for the Prevention of Post-endoscopic Retrograde Cholangiopancreatography Pancreatitis
Brief Title: Tailored Hydration for the Prevention of Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chonbuk National University Hospital (Other); Wonkwang University Hospital (Other); Kwangju christian hospital (Unknown); Presbyterian medical center (Unknown)
Responsible Party: Principal Investigator, Chang Hwan Park, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: CNUH-2018-080
Record Dates: First submitted 2018-06-03; First posted 2018-06-19 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Pancreatitis
Keywords: Endoscopic retrograde pancreatocholangiography; Pancreatitis; Lactate ringer's solution; Tailored therapy
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored standard hydration (Active Comparator): Patients will be randomly allocated to tailored standard hydration arm. Patients will receive hydration with lactated Ringer's solution with rate of 1.5 milliliter(mL)/kg/hr during and after ERCP. Hydration and feeding will be tailored by each patient's symptoms and serum amylase levels.
  Interventions: Drug: Tailored standard hydration
- Tailored aggressive hydration (Experimental): Patients will be randomly allocated to tailored aggressive hydration arm. Patients will receive hydration with lactated Ringer's solution with rate of 3.0 milliliter(mL)/kg/hr during and after ERCP and bolus injection of 20mL/kg over 1 hour after ERCP. Hydration and feeding will be tailored by each patient's symptoms and serum amylase levels.
  Interventions: Drug: Tailored aggressive hydration

INTERVENTIONS:
Drug: Tailored aggressive hydration — 1. Hydration with lactated Ringer's solution with rate of 3.0 milliliter(mL)/kg/hr during and after ERCP and bolus injection of 20mL/kg for 1 hour after ERCP.
  2. At 4 hours after ERCP (patients with ERPD stent insertion ; 6 hours), abdominal pain and serum amylase are checked. If pain (≥ Numeric rating scale (NRS) scale 3) is absent and amylase is below 1.5 times the upper normal limit (UNL), patient starts feeding and stops hydration. If patient has any of these signs, fasting and hydration continues.
  3. At 8 hours, if pain (<NRS scale 3) is absent, patient starts feeding and stops hydration. If patient has pain (≥ NRS scale 3) and previously checked amylase or re-checked serum amylase is above 3 times the UNL, patient is regarded as post-ERCP pancreatitis and receives 3mL/kg hydration. Patient with pain (≥ NRS scale 3) and previously checked serum amylase above 1.5 times but below 3 times the UNL, serum amylase is re-checked.
  Arms: Tailored aggressive hydration
Drug: Tailored standard hydration — 1. Hydration with lactated Ringer's solution with rate of 1.5milliliter(mL)/kg/hr during and after ERCP.
  2. At 4 hours after ERCP (patients with ERPD stent insertion ; 6 hours), abdominal pain and serum amylase are checked. If pain (≥ Numeric rating scale (NRS) scale 3) is absent and amylase is below 1.5 times the UNL(upper normal limit), patient starts feeding and stops hydration. If patient has any of these signs, fasting and hydration continues.
  3. At 8 hours, if pain (<NRS scale 3) is absent, patient starts feeding and stops hydration. If patient has pain (≥ NRS scale 3) and previously checked amylase or re-checked serum amylase is above 3 times the UNL, patient is regarded as post-ERCP pancreatitis and receives 3mL/kg hydration. Patient with pain (≥ NRS scale 3) and previously checked serum amylase above 1.5 times but below 3 times the UNL, serum amylase is re-checked.
  Arms: Tailored standard hydration

SUMMARY:
Aggressive hydration of lactated Ringer's solution has shown considerable beneficial effect in preventing post-ERCP(endoscopic retrograde cholangiopancreatography) pancreatitis. But the occurence rate of post-ERCP pancreatitis are near 10% and there are severe complications of aggressive hydration due to hypervolemia such pulmonary and peripheral edema, prolonged hospital stay and increased medical expense. Also there are no definite guidelines that suggest the duration and amount of hydration.

This study evaluates the efficacy and safety of tailored hydration depending on each patient's condition that indicates the likelihood of developing post-ERCP pancreatitis.

DETAILED DESCRIPTION:
ERCP(Endoscopic retrograde cholangiopancreatography) is the gold standard of diagnosis and treatment of pancreatobiliary disease. Pancreatitis is the most common complication after ERCP and can be lethally fatal.

The most fundamental modality of preventing and treatment of post-ERCP pancreatitis is hydration and recent studies showed considerable preventive effect of aggressive hydration of lactated Ringer's solution. Lactated Ringer's solution has very low risk of adverse reaction and low cost compared to other preventive modalities such as octreotide, corticosteroids and protease inhibitors.

Despite of these advantages of aggressive hydration of lactated Ringer's solution, the occurence rate of post-ERCP pancreatitis is near 10% and severe complications can develop due to hypervolemia caused by aggressive hydration such as pulmonary and peripheral edema, prolonged hospital stay and increased medical expense. Most of post-ERCP pancreatitis occur within several hours after ERCP and outpatients department based ERCP is suggested in some clinics by selecting patients with low risk of post-ERCP pancreatitis. A study compared the occurrence of post-ERCP pancreatitis between group with early feeding (4 hours after ERCP) and group with conventional feeding (24 hours after ERCP) and showed no difference. The most sensitive marker for predicting post-ERCP pancreatitis is abdominal pain and the occurrence time differs by whether endoscopic retrograde pancreatic duct (ERPD) stent insertion was performed or not. Patients without ERPD stent mostly develops abdominal pain at 2 hour after ERCP (0.5-2.5 hours) and patients with ERPD stent at 5 hour (0-68 hours). Also elevation of serum amylase level above 1.5 times the upper normal range after 4 hours of ERCP was suggested as useful marker for prediction of post-ERCP pancreatitis (AUROC 88.2%, 95% confidence interval 80.4%-90.6%).

The effectiveness of hydration for preventing post-ERCP pancreatitis is widely accepted but there are no definite guidelines that suggest the duration and amount of hydration.

Therefore, the purpose of this study is to evaluate the safety and efficacy of tailored hydration therapy based on markers that predicts the risk of post-ERCP pancreatitis development.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 20 years undergoing ERCP for the 1st time will be recruited

Exclusion Criteria:

* Age below 20 or above 80 years
* Underlying severe psychiatric illness
* Cardiac insufficiency (>New York Heart Association Class II heart failure)
* Renal insufficiency (eGFR <30mililiter/min/1.73m2)
* Respiratory insufficiency (defined as oxygen saturation < 90%)
* Poorly controlled blood sugar
* Ongoing hypotension including those with sepsis
* Ongoing acute pancreatitis
* Underlying disease of chronic pancreatitis
* Clinical signs of hypervolemia
* Hyponatremia (Na+ levels < 130 milliequivalent (mEq)/L))
* Hypernatremia (Na+ levels > 150mEq/L)
* Hyperkalemia (5.1 mEq/dL)
* Metabolic alkalosis
* Past history of endoscopic sphincterectomy or endoscopic papillary balloon dilatation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Development of post-ERCP pancreatitis | 24 hours
  Defined as pancreatic pain (≥ 3 on visual analogue numeric pain rating scale (0-10)) and serum amylase level 3 times the upper limit of normal.

SECONDARY OUTCOMES:
Clinical volume overload | 24 hours
  Defined by physical findings of peripheral edema and pulmonary rales
Hyperamylasemia | 24 hours
  Elevated serum amylase level above than upper limit of normal
Increased abdominal pain | 24 hours
  Defined as an increase in abdominal pain based on the visual analogue numeric pain rating score (0-10) following the ERCP compared to the score immediately prior to the ERCP.
Hospital stay | 1 year
  Whole duration of hospital admission days

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hwan Park, M.D, Ph.D, Study Director — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Anderson MA, Fisher L, Jain R, Evans JA, Appalaneni V, Ben-Menachem T, Cash BD, Decker GA, Early DS, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Ikenberry SO, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA. Complications of ERCP. Gastrointest Endosc. 2012 Mar;75(3):467-73. doi: 10.1016/j.gie.2011.07.010. No abstract available. PMID 22341094
- [Background] Buxbaum J, Yan A, Yeh K, Lane C, Nguyen N, Laine L. Aggressive hydration with lactated Ringer's solution reduces pancreatitis after endoscopic retrograde cholangiopancreatography. Clin Gastroenterol Hepatol. 2014 Feb;12(2):303-7.e1. doi: 10.1016/j.cgh.2013.07.026. Epub 2013 Aug 3. PMID 23920031
- [Background] Choi JH, Kim HJ, Lee BU, Kim TH, Song IH. Vigorous Periprocedural Hydration With Lactated Ringer's Solution Reduces the Risk of Pancreatitis After Retrograde Cholangiopancreatography in Hospitalized Patients. Clin Gastroenterol Hepatol. 2017 Jan;15(1):86-92.e1. doi: 10.1016/j.cgh.2016.06.007. Epub 2016 Jun 14. PMID 27311618
- [Background] Andriulli A, Leandro G, Federici T, Ippolito A, Forlano R, Iacobellis A, Annese V. Prophylactic administration of somatostatin or gabexate does not prevent pancreatitis after ERCP: an updated meta-analysis. Gastrointest Endosc. 2007 Apr;65(4):624-32. doi: 10.1016/j.gie.2006.10.030. PMID 17383459
- [Background] Rabago L, Guerra I, Moran M, Quintanilla E, Collado D, Chico I, Olivares A, Castro JL, Gea F. Is outpatient ERCP suitable, feasible, and safe? The experience of a Spanish community hospital. Surg Endosc. 2010 Jul;24(7):1701-6. doi: 10.1007/s00464-009-0832-5. Epub 2010 Jan 1. PMID 20044765
- [Background] Jeurnink SM, Poley JW, Steyerberg EW, Kuipers EJ, Siersema PD. ERCP as an outpatient treatment: a review. Gastrointest Endosc. 2008 Jul;68(1):118-23. doi: 10.1016/j.gie.2007.11.035. Epub 2008 Mar 4. PMID 18308308
- [Background] Park CH, Jung JH, Hyun B, Kan HJ, Lee J, Kae SH, Jang HJ, Koh DH, Choi MH, Chung MJ, Bang S, Park SW. Safety and efficacy of early feeding based on clinical assessment at 4 hours after ERCP: a prospective randomized controlled trial. Gastrointest Endosc. 2018 Apr;87(4):1040-1049.e1. doi: 10.1016/j.gie.2017.09.021. Epub 2017 Sep 28. PMID 28964747
- [Background] Kerdsirichairat T, Attam R, Arain M, Bakman Y, Radosevich D, Freeman M. Urgent ERCP with pancreatic stent placement or replacement for salvage of post-ERCP pancreatitis. Endoscopy. 2014 Dec;46(12):1085-94. doi: 10.1055/s-0034-1377750. Epub 2014 Sep 12. PMID 25216326
- [Derived] Cho E, Kim SH, Park CH, Yoon JH, Lee SO, Kim TH, Chon HK. Tailored Hydration With Lactated Ringer's Solution for Postendoscopic Retrograde Cholangiopancreatography Pancreatitis Prevention: A Randomized Controlled Trial. Am J Gastroenterol. 2024 Dec 1;119(12):2426-2435. doi: 10.14309/ajg.0000000000002903. Epub 2024 Jun 24. PMID 38912692